CLINICAL TRIAL: NCT02608073
Title: A Multi-Center Phase II Trial of Capecitabine (Xeloda) in Combination With Cisplatin as First Line Chemotherapy in Patients With Metastatic Nasopharyngeal Carcinoma
Brief Title: A Study of Capecitabine (Xeloda) as First-Line Chemotherapy in Participants With Metastatic Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18123
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Capecitabine; Cisplatin

ARMS (1):
- Capecitabine + Cisplatin (Experimental): Participants with metastatic nasopharyngeal cancer will receive combination treatment with capecitabine (1000 milligrams per meter square [mg/m^2] tablets twice daily [BID] orally) and cisplatin (100 mg/m^2/day intravenous [IV] infusion) for up to 8 cycles.
  Interventions: Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Capecitabine — Participants will receive oral capecitabine, 1000 mg/m^2 BID on Days 1 to 14 of each 21-day cycle, for up to 8 treatment cycles (24 weeks).
  Other Names: Xeloda
Drug: Cisplatin — Participants will receive cisplatin, 100 mg/m^2 via IV infusion on Day 1 of each 21-day cycle, for up to 8 treatment cycles (24 weeks).

SUMMARY:
This study will evaluate the efficacy, safety, tolerability, and effect on quality of life of oral capecitabine in combination with intravenous (IV) cisplatin in participants with metastatic nasopharyngeal cancer. Participants will receive up to 8 cycles of capecitabine treatment, and cisplatin will be administered on the first day of each cycle. The anticipated time on study treatment is up to 24 weeks, and the target sample size is 44 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 75 years of age
* Histologically confirmed, poorly differentiated or undifferentiated metastatic nasopharyngeal cancer with at least 1 measurable lesion which has not been irradiated
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Previous cytotoxic chemotherapy except adjuvant, concurrent, or neoadjuvant treatment completed at least 6 months before enrollment
* Clinically significant cardiac disease
* History of other malignancy within the last 5 years except cured basal cell cancer of the skin or cured cancer in situ of the cervix
* Radiotherapy within 4 weeks of treatment start or any prior radiotherapy performed to the indicator lesion(s) being measured in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 28 days after the last intake of study treatment (up to approximately 5 years)

SECONDARY OUTCOMES:
Overall survival | Up to approximately 18 months
Time to disease progression | Up to approximately 18 months
Duration of response | Up to approximately 18 months
Complete response rate | Up to approximately 18 months
Incidence of adverse events | Up to approximately 7 months
Quality of life according to Visual Analog Scale (VAS) score | Up to approximately 6 months
Treatment convenience/satisfaction according to VAS score | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Hong Kong, Hong Kong
- Yogyakarta, Indonesia
- Kuala Lumpur, Malaysia
- Taiwan (2):
  - Kueishan
  - Taipei
- Bangkok, Thailand